CLINICAL TRIAL: NCT03526146
Title: Preventing Loss of Independence Through Exercise (PLIÉ) in Persons With Mild Cognitive Impairment (MCI)
Acronym: MCI PLIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-23034
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Study participants will receive the PLIE intervention program (1 hour, 2 days/week, for 12 weeks) at the San Francisco VA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PLIE (Experimental): PLIE is an integrative exercise program that focuses on training procedural memory for the ability to perform the movements that are most needed for daily function (e.g., transitioning safely from sitting to standing) while increasing mindful body awareness and encouraging social connection. It combines elements from a wide range of Eastern and Western exercise modalities, including occupational therapy, physical therapy, yoga, tai chi, Feldenkrais, Rosen Method, dance movement therapy and mindfulness meditation.
  Interventions: Behavioral: Behavioral: Preventing Loss of Independence through Exercise (PLIE)

INTERVENTIONS:
Behavioral: Behavioral: Preventing Loss of Independence through Exercise (PLIE) — PLIE is an integrative exercise program that focuses on training procedural memory for the ability to perform the movements that are most needed for daily function (e.g., transitioning safely from sitting to standing) while increasing mindful body awareness and encouraging social connection. It combines elements from a wide range of Eastern and Western exercise modalities, including occupational therapy, physical therapy, yoga, tai chi, Feldenkrais, Rosen Method, dance movement therapy and mindfulness meditation.

SUMMARY:
Nearly 1 in 10 older Americans have dementia, which is a devastating condition that leads to a progressive loss of independence and functional status. Mild cognitive impairment (MCI) is an intermediate stage between the expected cognitive decline of normal aging and the more-serious decline of dementia. The investigators have developed a novel, integrative exercise program called Preventing Loss of Independence through Exercise (PLIE) that incorporates elements from Eastern and Western exercise modalities and is designed to build and maintain the capacity to perform basic functional movements while increasing mindful body awareness and enhancing social connection. Pilot study results suggest that PLIE is associated with meaningful improvements in physical function, cognitive function and quality of life in individuals with dementia, as well as reduced caregiver burden. The goal of the current study is to perform a randomized, controlled trial to test the efficacy of PLIE in older adults who have MCI but who do not yet have dementia. The investigators will also investigate the neural mechanisms underlying PLIE by acquiring brain imaging measures.

DETAILED DESCRIPTION:
The goal of the proposed study is to perform a randomized, controlled trial (RCT) to test the efficacy of a novel integrative exercise program called Preventing Loss of Independence through Exercise (PLIE) on function and quality of life in older adults living in the community with Mild cognitive impairment (MCI), which is an intermediate stage between the expected cognitive decline of normal aging and the more-serious decline of dementia.

Because current dementia medications have minimal impact on function and quality of life and do not stop or slow the disease course, it would be desirable if there were an intervention that could prevent or delay the onset of full-blown dementia. Moreover, there is growing evidence that behavioral interventions such as exercise have a variety of beneficial effects in individuals with dementia and MCI.

PLIE was developed based on recent discoveries in neuroscience and experimental psychology that have found that, although explicit memory (the ability to consciously recall new information) is impaired in individuals with dementia, implicit memory (unconscious learning that typically occurs through repeated exposure) is relatively preserved. Therefore, PLIE focuses on training procedural memory (unconscious learning of procedures) to build the strength and capacity to perform the movements that are most needed for daily function (e.g., transitioning safely from sitting to standing). In addition, to maximize the benefits of the training, PLIE integrates elements of Eastern and Western exercise modalities to develop mindful body awareness and enhance social connection.

The investigators have completed a pilot study of the PLIE program at an adult day center in San Francisco, CA. Results suggest that PLIE was associated with clinically meaningful improvements in cognitive function, physical performance and quality of life as well as reduced caregiver burden when compared with usual care at the facility. The current study will enable the investigators to build on this pilot study results by performing a RCT of PLIE for individuals who have MCI but who do not yet have dementia.

Study participants will be randomly assigned to receive the PLIE intervention program (1 hour, 2 days/week, 4 months) or Usual Care (UC) control (standard senior center activities, 1 hour, 2 days/week, 4 months) (N=40, 20/group) using a wait-list design. The co-primary outcomes are 4-month change in physical function (Short Physical Performance Battery, SPPB), cognitive function (Alzheimer's Disease Assessment Scale - cognitive subscale, ADAS-cog) and quality of life (Quality of Life in Alzheimer's Disease, QOL-AD). The investigators will also look at the 4-month change in the following neuroimaging measures: brain volume with structural magnetic resonance imaging (MRI), functional connectivity with resting-state functional MRI, cerebral perfusion with arterial-spin labeled MRI. To account for the wait-list design, all outcomes will be assessed at baseline, 4 months and 8 months.

The proposed project will address a critically important health problem related to optimizing functional status and quality of life in older individuals with MCI. The current study will utilize rigorous research methods to test the efficacy of an innovative and promising new program for older adults with MCI. If the program is successful, the investigators will work with VA and community-based organizations to implement PLIE more broadly.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Mild Cognitive Impairment (MCI) by primary care physician and/or neurologist
* English language fluency
* willing to attend PLIÉ classes 2 days/week
* ambulatory and able to take 2 steps without cane or walker; living in the community in a private home or apartment

Exclusion Criteria:

* Behavioral or physical issues that would be disruptive or dangerous to themselves or others (e.g., active psychosis, drug abuse, severe behavioral issues)
* Unable to attend 2 PLIÉ classes/week during the study period
* Physical or mental health condition that would make participation difficult (e.g., active psychosis, limited life expectancy)
* Contraindications to magnetic resonance imaging (MRI), including claustrophobia severe enough to prevent MRI examination, and presence of ferrometallic objects in the body that would interfere with MRI examination and/or cause a safety risk (e.g., pace makers, implanted stimulators, pumps).
* Started dementia medication (cholinesterase inhibitor or memantine) in past 3 months
* Planning to start/change any psychotropic medication during the study period
* Current participation in another research study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda I Chao, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barnes DE, Mehling W, Wu E, Beristianos M, Yaffe K, Skultety K, Chesney MA. Preventing loss of independence through exercise (PLIE): a pilot clinical trial in older adults with dementia. PLoS One. 2015 Feb 11;10(2):e0113367. doi: 10.1371/journal.pone.0113367. eCollection 2015. PMID 25671576
- [Result] Wu E, Barnes DE, Ackerman SL, Lee J, Chesney M, Mehling WE. Preventing Loss of Independence through Exercise (PLIE): qualitative analysis of a clinical trial in older adults with dementia. Aging Ment Health. 2015;19(4):353-62. doi: 10.1080/13607863.2014.935290. Epub 2014 Jul 14. PMID 25022459
- See also: Facebook page for PLIE program — https://www.facebook.com/plie4dementia
- See also: Osher Center description of PLIE program — http://www.osher.ucsf.edu/research/current-research/preventing-loss-of-independence-through-exercise-plie/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty-one (41) participants signed informed consent forms/were enrolled in the study. One participant did not meet study inclusion criteria; four participants withdrew for other reasons (e.g., time commitment/health issues, lack of interest); three participants were withdrawn after COVID-19 related shelter-in-place rules went into effect in San Francisco. Thirty-three(33) participants completed baseline assessments.
Period: Overall Study
Arm/Group | PLIE
Started | 33
Completed | 18
Not Completed | 15
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 6
Not completed — class canceled due to COVID-19 | 4

BASELINE CHARACTERISTICS:
Arm/Group | PLIE
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 25
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Alzheimer's Disease Assessment Scale-cognitive Subscale (ADAS-cog)
Description: The Alzheimer's Disease Assessment Scale - cognitive subscale (ADAS-cog) is one of the most commonly used outcome measures in dementia drug treatment trials and is one of the measures considered by the Food and Drug Administration for approval of dementia medications. It includes direct assessment of learning (10-word list), naming (objects), following commands, constructional praxis (figure copying), ideational praxis (mailing a letter), orientation (person, time, place), recognition memory and remembering test instructions. Scores may range from 0 to 70 with higher scores reflecting worse cognitive function. Prior studies have found the ADAS-cog to be valid and reliable with Cronbach's alpha greater than 0.8 and test-retest reliability above 0.9. Because we examined the difference from baseline to post-treatment, a positive change score indicates improvement while a negative change score indicates decline.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PLIE
Number analyzed (Participants) | 18
score on a scale | 2.83 (3.01)
Statistical Analysis 1: Comparison: PLIE; Test type: Superiority; p = 0.002, paired t-test

2. Secondary Outcome: Short Physical Performance Battery (SPPB)
Description: The SPPB was developed by the National Institute on Aging to provide an objective tool for measuring physical performance in older adults. Lower body strength is assessed based on time to complete 5 chair stands without using arms. Balance is assessed based on the ability to hold different stands for 10 seconds, including the side-by-side, semi-tandem and full tandem stands. Mobility is assessed based on usual walking speed over a 3-meter walking course. The total SPPB score is the sum of the 3 component scores and may range from 0 to 12. Higher scores reflect better performance. Because we examined the difference from baseline to post-treatment, a negative change score indicates improvement while a positive change score indicates decline.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PLIE
Number analyzed (Participants) | 18
score on a scale | -0.8 (1.7)
Statistical Analysis 1: Comparison: PLIE; Test type: Superiority; p = 0.047, paired t-test

3. Secondary Outcome: Interoceptive Self-Regulation, Assessed With the Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2)
Description: The MAIA is a 37-item self-report questionnaire, consists of eight scales: Noticing, Not-Distracting, Not-Worrying, Attention Regulation, Emotional Awareness, Interoceptive Self-Regulation, Body Listening, and Trust. To avoid overburdening participants with the entire questionnaire, we will focus on interoceptive self-regulation, the ability to regulate distress by attention to body sensations, which has previously been shown to respond to mindfulness interventions. Interoceptive Self-Regulation scores on the MAIA-2 range from 0-5, with lower scores indicating lower ability to regulate distress by paying attention to body sensations. Because we examined the difference from baseline to post-treatment, a negative change score indicates improvement while a positive change score indicates decline.
Time Frame: baseline to week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PLIE
Number analyzed (Participants) | 18
score on a scale | -0.8 (1.0)
Statistical Analysis 1: Comparison: PLIE; Test type: Superiority; p = 0.006, paired t-test

4. Secondary Outcome: Attention Regulation, Assessed With the Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2)
Description: The MAIA, a 37-item self-report questionnaire, consists of eight scales: Noticing, Not-Distracting, Not-Worrying, Attention Regulation, Emotional Awareness, Interoceptive Self-Regulation, Body Listening, and Trust. To avoid overburdening participants with the entire MAIA-2 questionnaire, we focused the ability to sustain and control attention to body sensations (i.e., attention regulation), which has been shown to respond to mindfulness interventions. Attention Regulation scores on the MAIA-2 range from 0-5, with lower scores indicating lower ability to sustain and control attention to body sensations. Because we examined change from baseline to post-treatment, a negative change score indicates improvement in the ability to sustain and control attention to body sensations.
Time Frame: baseline to week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PLIE
Number analyzed (Participants) | 18
score on a scale | -0.5 (0.9)
Statistical Analysis 1: Comparison: PLIE; Test type: Superiority; p = 0.05, paired t-test

5. Secondary Outcome: PROMIS Social Isolation
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Social Isolation questionnaire assesses perceptions of being avoided, excluded, detached, disconnected from, or unknown by, others with 4 questions (1- I feel left out; 2- I feel that people barely know me; 3- I feel isolated from others; 4-I feel that people are around me but not with me). Subjects respond to each statement with a Likert scale ranging from 1 (never) to 5 (always). Total scores range from 0-20, with higher scores indicating greater feelings of social isolation. Because we calculated a change score (baseline - post-treatment), a positive change score indicates a decrease in feelings of social isolation from baseline to post-treatment.
Time Frame: baseline to week 12
Population: Because this measure was not implemented at the beginning of the study, we do not have this measure for 6 study completers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PLIE
Number analyzed (Participants) | 12
score on a scale | 1.7 (1.8)
Statistical Analysis 1: Comparison: PLIE; Test type: Superiority; p = 0.009, paired t-test

ADVERSE EVENTS:
Time Frame: 12 weeks.
Description: PLIE creators attended classes.
Arm/Group | PLIE
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

LIMITATIONS AND CAVEATS:
We did not have an active control group. Therefore, we cannot rule out the possibility that practice, context, or placebo effects may have contributed to the behavioral findings and self report measures. Second, because the study only had one arm, the assessors were unblinded, which may have led to potential biases. A third limitation is that we performed numerous statistical tests without adjusting for multiple comparisons; therefore, there is a potential of false positives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT03526146/Prot_SAP_000.pdf